CLINICAL TRIAL: NCT03157336
Title: Toxicodietary and Genetic Determinants of Susceptibility to Neurodegeneration
Brief Title: Cassava Intervention Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Public Health, Democratic Republic of the Congo (Other Government)
Collaborators: National Institutes of Health (NIH) (NIH); Oregon Health and Science University (Other); Michigan State University (Other); University of Kinshasa (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Desire Tshala-Katumbay, Head Complex Morbidity Unit, Ministry of Public Health, Democratic Republic of the Congo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWA00017202; R01ES019841 (NIH)
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Neurotoxicity Syndrome, Cassava; Neurotoxicity Syndrome, Cyanate; Neurotoxicity Syndrome, Cyanide; Neurotoxicity Syndrome, Thiocyanate
Keywords: Cassava; Konzo; Cyanide; Cyanate; Thiocyanate; Carbamoylation; Isoprostanes; Oxidative Damage
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Intervention Model Description: We will implement a novel cassava processing method (wetting method, WTM) that safely removes cyanogenic compounds from cassava flour prior to human consumption in a stratified village-cluster randomized non-inferiority trial so as to compare the effectiveness of a peer-led intervention (Arm 1 = women training other women in the WTM) with that by community-health worker specialists (Arm 2= specialist led intervention arm)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-led Intervention (Experimental): Peers (community women in leading roles) training other women in the wetting method for safe processing of cassava in a non-inferiority intervention trial.
  Interventions: Other: Non Inferiority WTM Interventional Trial
- Specialist-led Intervention (Experimental): Specialists (nutritionists) training other women in the wetting method for safe processing of cassava in a non-inferiority intervention trial..
  Interventions: Other: Non Inferiority WTM Interventional Trial

INTERVENTIONS:
Other: Non Inferiority WTM Interventional Trial — The intervention will implement the WTM cassava processing technique in participating households. Twenty women (in leading roles) will be our principal candidates to serve as peer trainers. Together with a 20 community health worker specialists, these women will be trained in the WTM technique by the Kinshasa team of community health workers who are experts in the WTM method. Those who master the technique will then be certified as trainers to train and support other small groups of other mothers throughout a two-year period in the implementation of the WTM for the safer processing of food for their families. Both the community health worker specialists and trained women (prospective trainers) would have to be able to bring the cassava cyanogenic content to the lowest achievable level, which must be < 10 ppm as per the recommendations of the World Health Organization.

SUMMARY:
Investigators will implement a novel cassava processing method (wetting method, WTM) that safely removes cyanogenic compounds from cassava flour prior to human consumption in a stratified village-cluster randomized non-inferiority trial so as to compare the effectiveness of a peer-led intervention (women training other women in the WTM) with that by community-health worker specialists.

DETAILED DESCRIPTION:
The proposed project seeks methods to prevent and elucidate biomarkers of neurocognition and motor deficits associated with chronic dietary reliance on cyanogenic cassava, a staple food crop for more than 600 millions of people living in the tropics. Aim 1 will implement a novel cassava processing method (wetting method, WTM) that safely removes cyanogenic compounds from cassava flour prior to human consumption in a stratified village-cluster randomized non-inferiority trial so as to compare the effectiveness of a peer-led intervention (women training other women in the WTM) with that by community-health worker specialists (2 intervention training arms). Aim 2 will determine whether post-intervention reductions in cassava cyanogenic content and child U-SCN are associated with changes in biomarkers of cassava neurotoxicity particularly 8,12-iso-iPF2α-VI isoprostane (oxidant marker), carbamoylated albumin fragments KVPQVSTPTLVEVSR (residues 438-452) and LDELRDEGKASSAK (residues 206-219), or homocitrulline (carbamoylating markers), and scores at the KABC-II cognition and BOT-2 motor testing.

ELIGIBILITY:
Inclusion Criteria:

* Households with a konzo child and non-konzo sibling between 5 and 12 years
* Presence of a biological mother primarily responsible for the household food preparation and caring for the children
* Mother consenting to participate in this study

Exclusion Criteria:

* History of seizures
* History of cerebral malaria
* History of retroviral (HIV-HTLV) infections

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in food cyanogenic exposure | From baseline to 6-month time points
  Cassava cyanogenic content
Change in internal cyanogenic exposure | From baseline to 6-month time points
  Urinary concentrations of thiocyanate (U-SCN)
Change in oxidation damage | From baseline to 6-month time points
  Serum isoprostanes
Change in carbamoylation | From baseline to 6-month time points
  serum albumin peptidic carbamoylation
Change in carbamoylation surrogate | From baseline to 6-month time points
  serum homocitrulline

SECONDARY OUTCOMES:
Change in cognition performance | From baseline to 6-month time points
  Kaufman Assessment Battery for Children (KABC-II) for cognition testing score
Change in motor proficiency | From baseline to 6-month time points
  Motor proficiency Bruininks/Oseretsky Testing (BOT-2) score

CONTACTS AND LOCATIONS:
Overall Officials: Mumba Ngoyi, Study Director — Ministry of Health
Locations (1):
- INRB, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No